CLINICAL TRIAL: NCT00338962
Title: Naltrexone & SSRI in Alcoholics With Depression/PTSD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: HIC # 11637
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Alcoholism; Depression; PTSD
Keywords: SSRI; treatment; naltrexone; alcohol dependence; Desipramine; depression; PTSD
MeSH Terms: conditions — Alcoholism; Depression; Stress Disorders, Post-Traumatic | interventions — Paroxetine; Desipramine; Naltrexone; vivitrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Paroxetine and naltrexone (Active Comparator): Paroxetine was started at 10 mg per day and the dose was gradually increased over 2 weeks to 40 mg per day. Naltrexone was started at 25 mg the first day and 50 mg per day for the rest of the treatment.
  Interventions: Drug: paroxetine; Drug: Naltrexone
- paroxetine and placebo (Active Comparator): Paroxetine was started at 10 mg per day and the dose was gradually increased over 2 weeks to 40 mg per day.
  Interventions: Drug: paroxetine; Drug: Placebo
- Desipramine and naltrexone (Active Comparator): Desipramine was started at a dose of 25 mg per day. The dose was gradually increased over 2 weeks to 200 mg per day. Naltrexone was started at 25 mg the first day and 50 mg per day for the rest of the treatment.
  Interventions: Drug: desipramine; Drug: Naltrexone
- Desipramine and placebo (Active Comparator): Desipramine was started at a dose of 25 mg per day. The dose was gradually increased over 2 weeks to 200 mg per day.
  Interventions: Drug: desipramine; Drug: Placebo

INTERVENTIONS:
Drug: paroxetine — paroxetine (40mg/day)
  Other Names: paxil
  Arms: Paroxetine and naltrexone; paroxetine and placebo
Drug: desipramine — 200 mg per day
  Other Names: Norpramin
  Arms: Desipramine and naltrexone; Desipramine and placebo
Drug: Naltrexone — 50 mg per day
  Other Names: Vivitrol
  Arms: Desipramine and naltrexone; Paroxetine and naltrexone
Drug: Placebo — placebo
  Arms: Desipramine and placebo; paroxetine and placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of naltrexone in combination with an SSRI to reduce alcohol consumption in alcoholic patients with comorbid PTSD and depression.

We hypothesize that the combination of naltrexone and SSRI will exhibit a greater decrease in alcohol consumption than that seen with treatment with SSRI alone, or with a combination of another class of antidepressant and naltrexone. We also hypothesize that SSRI will be effective in treating PTSD and depressive symptoms and naltrexone will be well tolerated.

DETAILED DESCRIPTION:
OBJECTIVE: Alcoholics with current comorbid mental disorders constitute the majority of alcoholics in clinical settings. Although there are two FDA approved medications for the treatment of alcoholism (naltrexone and disulfiram), there are no established pharmacotherapies for individuals with comorbid alcoholism and psychiatric illnesses. Studies suggest that the class of antidepressants known as serotonin selective reuptake inhibitors (SSRIs) is effective in reducing alcohol use in depressed individuals. In addition, a small open label study has shown that SSRIs have similar effects on individuals with comorbid PTSD and alcoholism. Preclinical studies have shown that the combination of a serotonergic agent and naltrexone was more effective than either medication alone in suppressing alcohol intake. To address this issue, we are conducting a 13 week randomized clinical trial evaluating the effects of paroxetine, desipramine and naltrexone in reducing alcohol use in alcohol dependent individuals who currently meet DSM-IV diagnosis for Depressive Disorder or PTSD. RESEARCH PLAN: One hundred and twenty subjects who are alcohol dependent patients with comorbid PTSD or Depressive Disorder will be recruited from the following West Haven VA sources: the Substance Abuse Treatment program, the PTSD clinic, the Women's clinic, clinical referrals and advertisement. These subjects will be randomized in a double-blind fashion to one of four cells. We will compare paroxetine versus desipramine and naltrexone versus placebo. The antidepressant will be started at a low dose and titrated upward on a fixed schedule. The target dose will be 40mg for paroxetine and 200mg for desipramine. Minimum dosage permitted for study retention will be 20mg for paroxetine and 150mg for desipramine. Pharmacological treatments will last 13 weeks. Psychosocial treatment will involve medication compliance therapy, using the Microelectric Event Monitoring (MEMS) bottle caps. The specific aim of the research is to compare the relative effectiveness of paroxetine versus desipramine and naltrexone versus placebo in reducing the quantity and frequency of alcohol consumption. METHODOLOGY: The primary outcome measures of major interest will include: frequency and quantity of alcohol consumption, self-reported craving, self-reported psychiatric and emotional distress, diagnostic assessment or psychiatric symptoms and side effects. These outcomes will be measured by the following: self-assessments, Timeline Followback, Hamilton Depression and anxiety scales, CAPS, ASI, Quality of Life, breathalyzer tests and monthly liver function tests.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of alcohol dependence and current DSM-IV depressive disorder or PTSD
* a recent episode of heavy drinking
* outpatient, sober from alcohol and other abused substance for at least 2 days before randomization
* stable medication regiment for at least 2 weeks
* women on adequate methods of contraception

Exclusion Criteria:

* current opioid dependence or abuse
* history (within the last 3 months) of opioid dependence or abuse
* pregnant
* history of psychotic disorders or current treatment with antipsychotic medications
* medication thought to influence drinking including: acamprosate, disulfiram, naltrexone, ondansetron, valproic acid or tegretol
* current (within the lst 6 months) use of MAO inhibitors
* suicidal active ideation or intent
* significant underlying medical condition
* history of cardiac condition abnormalities

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2001-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ismene Petrakis, M.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare Systems, West Haven, Connecticut, United States

REFERENCES:
- [Derived] Petrakis IL, Ralevski E, Desai N, Trevisan L, Gueorguieva R, Rounsaville B, Krystal JH. Noradrenergic vs serotonergic antidepressant with or without naltrexone for veterans with PTSD and comorbid alcohol dependence. Neuropsychopharmacology. 2012 Mar;37(4):996-1004. doi: 10.1038/npp.2011.283. Epub 2011 Nov 16. PMID 22089316
- See also: Published paper — http://www.ncbi.nlm.nih.gov/pubmed/22089316

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paroxetine and Naltrexone | Paroxetine and Placebo | Desipramine and Naltrexone | Desipramine and Placebo
Started | 22 | 20 | 22 | 24
Completed | 14 | 16 | 16 | 21
Not Completed | 8 | 4 | 6 | 3
Not completed — Lost to Follow-up | 3 | 3 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — No Transportation | 2 | 0 | 0 | 0
Not completed — Time Constraint | 2 | 0 | 0 | 0
Not completed — Moved | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Poor Compliance | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paroxetine and Naltrexone | Paroxetine and Placebo | Desipramine and Naltrexone | Desipramine and Placebo | Total
Number analyzed (Participants) | 22 | 20 | 22 | 24 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.14 (6.71) | 49.15 (8.95) | 47.05 (9.96) | 47.04 (9.72) | 47.1 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 4 | 3 | 8
  Male | 22 | 19 | 18 | 21 | 80

OUTCOME MEASURES:

1. Primary Outcome: Mean Self-report Weekly Craving Via Obsessive Compulsive Drinking Scale (OCDS)
Description: The OCDS is a 14-item (rated 0-4), self-administered questionnaire for characterizing and quantifying the obsessive and compulsive cognitive aspects of craving and heavy (alcoholic) drinking, such as drinking-related thought, urges to drink, and the ability to resist those thoughts and urges. A higher total score indicates higher craving and ranges from 0-48.
Time Frame: beginning of treatment (week 1), and end of treatment (13 weeks)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Paroxetine and Naltrexone | Paroxetine and Placebo | Desipramine and Naltrexone | Desipramine and Placebo
Number analyzed (Participants) | 14 | 16 | 16 | 21
units on a scale
  Week 1 | 21.273 (2.547) | 20.700 (2.672) | 18.500 (2.547) | 21.458 (2.439)
  Week 13 | 10.013 (3.009) | 9.690 (3.025) | 4.296 (2.847) | 7.489 (2.483)

2. Primary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: The CAPS is the gold standard in PTSD assessment. The CAPS-5 is a 30-item structured interview that can be used to:
  Make current (past month) diagnosis of PTSD Make lifetime diagnosis of PTSD Assess PTSD symptoms over the past week Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). A higher score is associated with higher severity of PTSD. The score is interpreted as follows: 0-19=Asymptomatic/few symptoms 20-39=Sub-threshold/mild PTSD 40-59=Threshold PTSD/moderate 60-79=Severe PTSD >80=Extreme PTSD
Time Frame: beginning of treatment (week 1), and end of treatment (13 weeks)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Paroxetine and Naltrexone | Paroxetine and Placebo | Desipramine and Naltrexone | Desipramine and Placebo
Number analyzed (Participants) | 14 | 16 | 16 | 21
units on a scale
  Beginning of Treatment | 73.54 (5.007) | 69.810 (5.166) | 62.500 (5.047) | 77.833 (4.832)
  End of Treatment | 40.024 (5.53) | 36.591 (5.570) | 26.751 (5.353) | 41.392 (4.949)
Statistical Analysis 1: Comparison: Paroxetine and Naltrexone vs Paroxetine and Placebo vs Desipramine and Naltrexone vs Desipramine and Placebo; Test type: Superiority or Other; p = 0.00, Mixed Models Analysis — Bonferonni adjustments were applied. Mixed effects models were used to assess changes in PTSD symptoms over time; F=49.633

3. Primary Outcome: Hamilton Depression Rating Scale (HAM-D)
Description: The HAM-D ranges from 0 (Normal) to >23 (Very Severe Depression)
Time Frame: beginning of treatment (week 1), and end of treatment (13 weeks)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Paroxetine and Naltrexone | Paroxetine and Placebo | Desipramine and Naltrexone | Desipramine and Placebo
Number analyzed (Participants) | 14 | 16 | 16 | 21
units on a scale
  Beginning of Treatment | 13.273 (1.112) | 10.950 (1.167) | 11.195 (1.132) | 13.167 (1.065)
  End of Treatment | 9.328 (1.256) | 8.238 (1.299) | 8.563 (1.201) | 8.943 (1.117)

4. Primary Outcome: Mean Number of Side Effects
Description: Differences in mean number of side effects reported for each group. Side effects and common adverse symptoms were evaluated by the research staff weekly, using a modified version of the ystematic Assessment for Treatment Emergent Events. The symptoms that are known to be associated with treatment with desipramine, paroxetine, and naltrexone were specifically screened or on a weekly basis. The symptoms were then clustered into the following categories: gastrointestinal, emotional, cold and flu symptoms, skin, sexual, neurological, and cardiac.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: side effects
Arm/Group | Paroxetine and Naltrexone | Paroxetine and Placebo | Desipramine and Naltrexone | Desipramine and Placebo
Number analyzed (Participants) | 22 | 20 | 22 | 24
side effects
  Gastrointestinal symptoms | 3.651 (.487) | 2.688 (.513) | 3.052 (.475) | 3.653 (.431)
  Emotional Symptoms | 4.874 (.686) | 3.963 (.719) | 3.727 (.689) | 5.248 (.629)
  Neurological Symptoms | 6.212 (1.058) | 5.078 (1.106) | 4.201 (1.047) | 4.566 (.970)
  Cold Symptoms | 2.182 (.490) | 2.393 (.512) | 1.891 (.483) | 2.253 (.447)
  Skin Symptoms | 1.002 (.240) | .859 (.252) | .591 (.236) | 1.057 (.215)
  Sexual Symptoms | .877 (.241) | .932 (.252) | .737 (.238) | .736 (.219)
  Cardiac Symptoms | .416 (.093) | .474 (.101) | .389 (.089) | .356 (.076)
Statistical Analysis 1: Comparison: Paroxetine and Naltrexone vs Paroxetine and Placebo vs Desipramine and Naltrexone vs Desipramine and Placebo; Gastrointestinal symptoms compared; Test type: Superiority or Other; p = 0.007, ANOVA

ADVERSE EVENTS:
Time Frame: 9 weeks afters study medication
Arm/Group | Paroxetine and Naltrexone | Paroxetine and Placebo | Desipramine and Naltrexone | Desipramine and Placebo
Serious Adverse Events (participants affected / at risk) | 1/22 | 2/20 | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 1/22 | 1/20 | 2/22 | 2/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxetine and Naltrexone (N=22) | Paroxetine and Placebo (N=20) | Desipramine and Naltrexone (N=22) | Desipramine and Placebo (N=24)
Death (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Subject was injured at work. Death was not study related.
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Hospitalized for severe anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paroxetine and Naltrexone (N=22) | Paroxetine and Placebo (N=20) | Desipramine and Naltrexone (N=22) | Desipramine and Placebo (N=24)
Dizziness and Lightheadedness (Nervous system disorders) | 0 | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Incarcerated for intoxication (General disorders) | 1 | 0 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 — 9 weeks after discontinuing meds

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes